CLINICAL TRIAL: NCT00267891
Title: Changes in Activation Patterns in the Ventro-Medial Prefrontal Cortex of Healthy Adolescents During the Imagination and Observation of Aggressive Behavior
Brief Title: Brain Changes in Adolescents While Imagining and Observing Aggressive Behavior
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060048; 06-N-0048
Record Dates: First submitted 2005-12-21; First posted 2005-12-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-08-12

CONDITIONS: Aggressive Behavior
Keywords: Healthy Control Subjects; Aggression; Prefrontal Cortex Function; Children and Adolescents; Healthy Volunteer; HV
MeSH Terms: conditions — Aggression

SUMMARY:
This study will use functional magnetic resonance imaging (fMRI) to examine what happens in the brains of adolescents when they are exposed to violent media and how imagining aggressive behavior affects brain function. The study will measure physiological changes (such as the amount of electricity generated by the skin, heart rate, and breathing rate) related to these tasks during fMRI. MRI uses a magnetic field and radio waves to obtain images of body organs and tissues. For fMRI, the subject performs certain tasks during the MRI scanning to examine changes in the brain regions that are involved with those tasks. During the scan, the subject lies in a metal cylinder (the scanner), wearing earplugs to muffle loud noises that occur with the scanning.

Healthy right-handed native English-speaking males between 14 and 17 years of age may be eligible for this study. Candidates are screened with a neurological examination and neuropsychological testing that includes questions about their feelings, experiences, and behavior, and tests of reading level and intelligence.

Participants undergo fMRI and fill out questionnaires before and after the scanning. Some children are asked to play 20 minutes of video games before the test. During the scan, the child views short neutral video clips and video clips of people fighting or imagine self-defense situations. The child is asked to rate the video clips for their aggressive content or tell how he or she feels about the imagined situations. Two small straps are wrapped around the child's index and middle fingers to measure changes in the amount of electricity generated by the skin, and a strap at the ring finger measures the child's heart rate. A band around the child's chest records breathing rates.

Children who cannot or do not want to undergo MRI testing may be asked to view commercially available video clips of people fighting and neutral video scenes, such as sports scenes. They are asked to rate them on their violent content and excitement, or to rate the video games they have played on their violent/nonviolent content and their popularity. In addition, the children fill out questionnaires about their media use and exposure to violence.

All participating families are contacted by telephone 1 day and 2 weeks after the experiment for parents to answer questions about how the child has been doing and for the children to answer questions about their feelings.

DETAILED DESCRIPTION:
Objective. The purpose of the protocol is to localize the prefrontal cortical regions mediating aggressive behavior. Utilizing two different experimental neuropsychological tasks during functional MRI, we will investigate hypotheses regarding the role of the ventro-medial prefrontal cortex in processing imagined and observed aggressive behavior. Additionally, we will determine the relationship between non-frontal neural structures involved in emotional expression, such as the amygdala, and the prefrontal structures involved in executive functions that may modulate aggressive behavior. We will record skin conductance responses (SCRs), heart rates, and respiration during the experiments to investigate autonomic changes during the processing of aggressive behavior.

Study Population. In three separate studies, normal adolescent volunteers will participate in experiments dealing with processing of aggressive behavior using functional magnetic resonance imaging (fMRI). In addition, we will conduct two pre-studies in normal adolescent volunteers in order to determine appropriate stimuli for the fMRI studies.

Design. The experiments we are conducting will employ within-subject, rapid event-related fMRI designs to determine whether the observation and imagination of aggressive behavior deactivates the ventro-medial prefrontal cortex (VM-PFC) and how varying intensities of imagined and observed aggressive acts may influence changes in activation patterns in the VM-PFC.

Outcome Measures. The data collected will consist of fMRI activation images corresponding to varying intensities of observed or imagined aggression, questionnaire results, amplitudes of the skin conductance responses, heart rates, and respiration parameters. The results gained from this protocol will provide further evidence for the role of the ventro-medial prefrontal cortex in processing aggressive behavior, particularly in adolescents.

ELIGIBILITY:
* INCLUSION CRITERIA:

In all the studies, participants will consist of male adolescent healthy, native English-speaking, right-handed volunteers. Participants will range in age from 14 to 17 years old and they will be included regardless of race.

EXCLUSION CRITERIA:

Non-native English speakers and non-right handers will be excluded, as will non-neurologically normal volunteers. Subjects younger than 14 and older than 17 years of age will be excluded.

Subjects with any of the following will be excluded from MRI testing: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body, such as metal shavings; permanent eyeliner; insulin pump; or irremovable body piercing will be excluded from the study due to the possible dangerous effects of the magnet upon metal objects in the body.

Individuals with a neurological or psychiatric history, including significant aggressive behavior and drug abuse, or with a medical condition that would compromise our interpretation of the fMRI results will be excluded. Adolescents with attentional, cognitive, or learning difficulties or impairments cannot take part in the study. An intelligence quotient less then 80 will be exclusion criteria for this study. Individuals with a current or past history of post-traumatic stress disorder or other psychiatric disorders or individuals with a history of physical or sexual abuse will be excluded as they may be disturbed by the exposure to violent stimuli. Furthermore, we will exclude adolescents who take centrally acting medications. The presence or absence of these conditions will be determined by a standardized neuropsychiatric interview, questionnaires, ability testing, and standard phone or in-person intake (see screening section).

Adolescents who have been trained in martial arts will be excluded from our studies.

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2005-12-14; Study Completion 2010-08-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anderson CA, Bushman BJ. Effects of violent video games on aggressive behavior, aggressive cognition, aggressive affect, physiological arousal, and prosocial behavior: a meta-analytic review of the scientific literature. Psychol Sci. 2001 Sep;12(5):353-9. doi: 10.1111/1467-9280.00366. PMID 11554666
- [Background] Anderson CA, Dill KE. Video games and aggressive thoughts, feelings, and behavior in the laboratory and in life. J Pers Soc Psychol. 2000 Apr;78(4):772-90. doi: 10.1037//0022-3514.78.4.772. PMID 10794380
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.